CLINICAL TRIAL: NCT02504333
Title: A Phase I/II Study of Nab-paclitaxel (Abraxane) and Gemcitabine Followed by Modified FOLFOX (AG-mFOLFOX) in Patients With Previously Untreated, Metastatic Pancreatic Adenocarcinoma
Brief Title: Phase I/II Study of Nab-paclitaxel and Gemcitabine Followed by AG-mFOLFOX in Patients With Metastatic Pancreatic Adenocarcinoma
Acronym: SEQUENCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Spanish Cooperative Group for the Treatment of Digestive Tumours (TTD) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TTD-14-05
Record Dates: First submitted 2015-07-20; First posted 2015-07-21 (Estimated); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Metastatic Pancreatic Adenocarcinoma
Keywords: metastatic pancreatic adenocarcinoma; Nab-paclitaxel; Gemcitabine; modified FOLFOX
MeSH Terms: interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AG (Active Comparator): nab-Paclitaxel followed by Gemcitabine
  Interventions: Drug: nab-paclitaxel; Drug: gemcitabine
- AG-mFOLFOX (Experimental): nab-Paclitaxel followed by Gemcitabine and FOLFOXm at dose levels selected from the phase I trial
  Interventions: Drug: m-FOLFOX; Drug: nab-paclitaxel; Drug: gemcitabine

INTERVENTIONS:
Drug: nab-paclitaxel — Day 1-8-15: Intravenous, 125 mg/m2 over 30 minutes
  Arms: AG
Drug: gemcitabine — Day 1-8-15: Intravenous, 1.000 mg/m2 over 30 minutes
  Arms: AG
Drug: m-FOLFOX — Day 28 according to the dose levels stablished in Phase I
  Arms: AG-mFOLFOX
Drug: nab-paclitaxel — Day 1-8-15: Intravenous 30 minutes according to the dose levels stablished in Phase I
  Arms: AG-mFOLFOX
Drug: gemcitabine — Day 1-8-15: Intravenous 30 minutes according to the dose levels stablished in Phase I
  Arms: AG-mFOLFOX

SUMMARY:
The purpose of this study is to assess the safety and efficacy of nab-paclitaxel (Abraxane) and gemcitabine followed by modified FOLFOX (AG-mFOLFOX) in patients with previously untreated, metastatic pancreatic adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed pancreatic adenocarcinoma
2. Stage IV disease (metastatic only)
3. No prior systemic therapy for their diagnosis (except in adjuvant/neoadjuvant setting>six months previously)
4. ECOG performance status of 0-1
5. At least 18 years of age
6. Evidence of either or both of the following RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥10 mm with spiral CT scan)
7. Female patients must be either surgically sterile or postmenopausal, or if of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment and agree to use effective barrier contraception during the period of therapy. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy. The definition of effective contraception will be based on the judgment of the investigator.
8. Adequate bone marrow function:

   * ANC ≥ 1500/uL
   * platelet count ≥ 100,000/uL
   * hemoglobin ≥ 9.0 g/dL
9. Adequate hepatic function:

   * Total bilirubin ≤ 1.5 X ULN
   * AST (SGOT) ≤ 2.5 X ULN
   * ALT (SGPT) ≤ 2.5 X ULN
10. Adequate renal function as determined by either:

    - Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used).
11. Ability to understand the nature of this study protocol and give written informed consent.
12. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.

Exclusion Criteria:

1. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that, in the opinion of the investigator, renders the subject at high risk from treatment complications or might affect the interpretation of the results of the study.
2. Presence of central nervous system or brain metastases.
3. Life expectancy < 12 weeks
4. Pregnancy (positive pregnancy test) or lactation.
5. Pre-existing sensory neuropathy > grade 1.
6. Clinically significant cardiac disease (e.g. congestive heart failure, symptomatic coronary artery disease and cardiac arrhythmias not well controlled with medication) or myocardial infarction within the last 12 months.
7. Major surgery and/or radiotherapy within 4 weeks of the start of study treatment, without complete recovery.
8. Prior malignancy except for adequately treated basal cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other form of cancer from which the patient has been disease-free for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2015-07; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity for the AG-mFOLFOX combination | 12 weeks
  Primary outcome phase I.
Rate of overall survival al 12 months | 12 weeks
  Primary outcome phase II

SECONDARY OUTCOMES:
Rate of overall survival at 6 months | 54 months
Rate of overall survival at 24 months | 54 months
Time to tumor progression | 54 months
Progression free survival | 54 months
Overall Survival | 54 months
Objective radiographic response | 54 months
  Secondary outcome Phase I and Phase II
CA 19-9 biomarker response | 54 months
Safety profile of this combination (AG-mFOLFOX) using NCI-CTCAE v.4 criteria | 54 months
  Secondary outcome Phase I and Phase II
To assess the Quality of Life of the patients through the EORTC QLQ-C30/PAN26 and EORTC QLQ-CIPN20 questionnaires | 54 months
  Secondary outcome Phase I and Phase II

OTHER OUTCOMES:
microRNA expression levels and their correlation with tumour-efficacy parameters | 54 months
Biomarker determination (tissue sample at basal point and blood samples at basal and at the end of treatment). Correlation with treatment response | 54 months

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Carrato, MD PhD, Study Chair — Hospital Universitario Ramón y Cajal; Carmen Guillén, MD, Study Chair — Hospital Universitario Ramón y Cajal
Locations (1):
- Spanish Cooperative for Digestive Tumour Therapy (TTD), Madrid, Spain

REFERENCES:
- [Derived] Carrato A, Pazo-Cid R, Macarulla T, Gallego J, Jimenez-Fonseca P, Rivera F, Cano MT, Rodriguez-Garrote M, Pericay C, Ales I, Layos L, Grana B, Iranzo V, Gallego I, Garcia-Carbonero R, de Mena IR, Guillen-Ponce C, Aranda E. Nab-Paclitaxel plus Gemcitabine and FOLFOX in Metastatic Pancreatic Cancer. NEJM Evid. 2024 Feb;3(2):EVIDoa2300144. doi: 10.1056/EVIDoa2300144. Epub 2024 Jan 23. PMID 38320486
- See also: Related Info — http://www.ttdgroup.org